CLINICAL TRIAL: NCT02605330
Title: Kinetics of Plasma Fibrinogen During Cardiac and Thoracic Aortic Surgery
Brief Title: Kinetics of Plasma Fibrinogen in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 193/15
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Fibrinogens, Abnormal
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood containing all components
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fibrinogen plasma level in CABG: In all patients undergoing coronary artery bypass grafting (CABG) the investigators plan to measure the fibrinogen plasma level
  Interventions: Procedure: Fibrinogen plasma level
- Fibrinogen plasma level in AVR: In all patients undergoing aortic valve replacement (AVR) the investigators plan to measure the fibrinogen plasma level
  Interventions: Procedure: Fibrinogen plasma level
- Fibrinogen plasma level in AAR: In all patients undergoing aortic arch replacement (AAR) the investigators plan to measure the fibrinogen plasma level
  Interventions: Procedure: Fibrinogen plasma level

INTERVENTIONS:
Procedure: Fibrinogen plasma level — At 12 different time points investigators plan to measure the plasma fibrinogen level with conventional coagulation tests (Clauss fibrinogen) and with ROTEM.

SUMMARY:
The study intends to measure fibrinogen plasma levels during the first 24 hrs in cardiac and thoracic surgical patients who undergo surgical procedures using extracorporeal circulation.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients undergoing coronary artery bypass grafting, aortic valve replacement or thoracic aortic surgery
* Signed written informed consent

Exclusion Criteria:

* Participation in another study
* Language barrier to understand study purposes (e.g. french as a native language)
* Preoperative low level of plasma fibrinogen (< 1.75 g/l)
* Preoperative anemia (Hb < 10g/dl)
* Emergency treatment
* Intake of anticoagulants other than aspirin within 14 days preceding surgery.
* Known coagulation disorder.
* Jehovah's witnesses

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with extracorporeal bypass
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Plasma fibrinogen concentration | through study completion, an average of 1 year
  Conventional (Clauss) and thromboelastometric measurement (FIBTEM)

SECONDARY OUTCOMES:
Periprocedural thromboembolic complications | through study completion, an average of 1 year
Thoracic drain loss | through study completion, an average of 1 year
  Measurement of the amount of blood collected by the thoracic drain (ml)
In-hospital mortality | through study completion, an average of 1 year
Intensive Care Unit (ICU) length of stay | through study completion, an average of 1 year
Platelet count | through study completion, an average of 1 year
  Measurement of platelet count in the laboratory
Prothrombin time (Quick) | through study completion, an average of 1 year
  Measurement of Quick in the laboratory
Activated partial thromboplastin time (aPTT) | through study completion, an average of 1 year
  Measurement of aPTT in the laboratory
Thromboelastometric (ROTEM) parameters (e.g., INTEM, EXTEM, HEPTEM) | through study completion, an average of 1 year
  Measurement of ROTEM parameter (unit mm) in the laboratory
Thrombin concentration | through study completion, an average of 1 year
  Thrombin concentration in the plasma as measured in the laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland